CLINICAL TRIAL: NCT05597072
Title: Infection Control - Time-dependant Bacterial Air Contamination in the Operating Room
Brief Title: Bacterial Air Contamination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Camilla Wistrand (Other)
Responsible Party: Sponsor-Investigator, Camilla Wistrand, University Hospital in Örebro, Örebro University, Sweden
Organization: Örebro University, Sweden (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: BAirCon 2022
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Infection Control
Keywords: Infection control
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the evening before an elective surgery the sterile surgical goods will be prepared under calm circumstances with only 2 persons in the OR (intervention). Thereafter, the sterile goods will be protected with sterile covers and time pending surgery will be approximately 12 hours (intervention).
  Interventions: Behavioral: Intervention
- Control (Active Comparator): The control is to prepare the sterile goods in the morning with more people in the OR (approximately 4-5 persons).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Less people within the OR but longer waiting time.
  Arms: Intervention
Behavioral: Control — More people in the OR but shorter waiting time
  Arms: Control

SUMMARY:
Aim is to compare the effect of number of persons and time-dependant bacterial air contamination on sterile goods, using different preparation conditions and protective sterile covers.

Research questions Is there a difference in bacterial air contamination during preparation of the sterile surgical goods with 2 persons (intervention) compared with 4-5 persons (control) in the OR? Is there a time-dependent difference in bacterial air contamination pending surgery for 1 hour (control) compared to approximately 12 hours (intervention) when the sterile goods are protected with sterile covers? Is there a time-dependent difference in bacterial air contamination pending surgery if sterile goods are protected or not, by sterile covers? Is there any differences in surgical site infections between the groups? What type of bacteria contain the air contamination? Is there antibiotic resistant bacterial air contamination?

DETAILED DESCRIPTION:
Intervention - In the evening before an elective surgery the sterile surgical goods will be prepared under calm circumstances with only 2 persons in the OR (intervention). Thereafter, the sterile goods will be protected with sterile covers and time pending surgery will be approximately 12 hours (intervention). The control is to prepare the sterile goods in the morning with more people in the OR (approximately 4-5 persons). Thereafter, the sterile goods will be protected with sterile covers (time pending surgery will be approximately one hour). For allocation, a computer-generated randomization list will be produced and an independent secretary will be arranging the printed notes showing the group assignment in ordered, sealed, non-transparent envelopes.

To measure the time pending surgery tables will be arrange with blood agar plates to measure the bacterial air contamination. There will be two tables, one protected with sterile covers and one left without protective covers (in both intervention- and control group).

Outcomes and materials - Primary outcome is bacterial growth isolated by aerobe and anaerobe blood agar plates (haematin agar medium 4.3% w/v [Colombia Blood Agar Base] supplemented with 6% w/v chocolatized defibrinated horse blood) and FAA plates (LAB 90 Fastidious Anaerobe Agar 4.6% w/v supplemented with 5% w/v defibrinated horse blood). Secondary outcome is surgical site infections with comparison of bacteria type.

Data collection - A total of 1260 blood agar plates will be used to capture bacterial air contamination. To capture differences in bacterial air contamination during different preparation conditions of the sterile goods, six agar plates (three haematin and three FAA) will be set on a table as the preparation begins. When preparation is complete the agar plates will be collected, by closing the lid of the agar plates. To measure the time-dependant bacterial air contamination pending surgery new agar plates (three haematin and three FAA) which will be set on tables for both intervention- and control group and covered with sterile drapes. To measure the effectiveness of sterile coverage from bacterial air contamination agar plates will be left uncovered pending surgery in both intervention- and control group. When preparing the patient for surgery the covers will be removed and all the plates will be collected by closing the lids.

Microbiology - The plates will be analysed at the Department of Laboratory Medicine, Clinical Microbiology, Örebro University Hospital, according to a specific study protocol. The haematin plates will be incubated at 36°C under aerobic conditions while the FAA plates will be incubated under anaerobic conditions (10% H2, 10% CO2, 80% N2) at 37°C. After 24 and 48 h of aerobic incubation and five days of anaerobic incubation, bacterial growth will be determined quantitatively by counting colony-forming units per plate. The isolates will be identified by routine diagnostic procedures and determined to species level via matrix-assisted laser desorption/ionization time-of-flight mass spectrometry (Microflex LT and Biotyper 3.1, Bruker Daltonik, Bremen, Germany).

Standard antibiotic susceptibility testing for staphylococci will be performed by the disc diffusion test for cefoxitin (30 mg), fusidic acid (10 mg), erythromycin (15 mg), clindamycin (2 mg), trimethoprim/sulfamethoxazole (25 mg), gentamicin (10 mg), norfloxacin (10 mg), ciprofloxacin (5 mg), and rifampin (5 mg) (all antibiotic discs from Oxoid, Basingstoke, UK) with a 0.5 McFarland bacterial suspension in 0.85% NaCl on Mueller-Hinton II agar 3.8% w/v plates (BD Diagnostic Systems, Sparks, MD, USA). After 16-20 h of incubation at 35°C, the zone diameters will be measured and each isolate will be evaluated according to European Committee on Antimicrobial Susceptibility Testing breakpoints (http://www.eucast.org). Isolates resistant to at least three of the antibiotic groups tested will be considered multidrug resistant.

The susceptibility of Cutibacterium acnes to benzylpenicillin and clindamycin will be investigated using a gradient test. Minimum inhibitory concentrations will be determined by Etest (bioMe´rieux, Marcy l'Etoile, France) on FAA plates (LAB M) with 0.5 McFarland suspensions of bacteria in NaCl and incubation at 36°C in an anaerobic atmosphere for 24 h. For metronidazole, a disc (Oxoid) will be used. Bacterial genomic sequencing may be analysed in order to understand if the bacteria derives from the persons within the OR or the hospital environment.

All data regarding postoperative infections will be retrieved from a local register Carath, Department of Cardiothoracic and Vascular surgery. A case report form (CRF) will be used to collect data regarding patient characteristics, OR settings (e.g. temperature, air humidity, number of persons, number of door openings) and surgical data (e.g. type of surgery, time for surgery).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (n=70) undergoing cardiac surgery at the Department of Cardiothoracic and Vascular Surgery at Örebro University Hospital (ÖUH), Region Örebro County will be identified. Inclusion criteria: patients undergoing cardiac surgery by median sternotomy; coronary artery bypass grafting (CABG), aneurysm, valve replacement or combination surgery.

Exclusion Criteria:

* Patients where partial thoracotomy or endovascular procedures are performed. Patients with infection and procedures as infective endocarditis. No research nurse available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Colony forming units | from one to 15 hours
  Bacterial growth

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Wistrand, PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wistrand C, Soderquist B, Sundqvist AS. The effect of five versus two personnel on bacterial air contamination during preparation of sterile surgical goods in the operating room: a randomised controlled trial. Antimicrob Resist Infect Control. 2025 Jun 15;14(1):68. doi: 10.1186/s13756-025-01589-4. PMID 40518530
- [Derived] Wistrand C, Soderquist B, Friberg O, Sundqvist AS. Bacterial air contamination and the protective effect of coverage for sterile surgical goods: A randomized controlled trial. Am J Infect Control. 2025 Apr;53(4):467-472. doi: 10.1016/j.ajic.2024.12.012. Epub 2024 Dec 16. PMID 39694445